CLINICAL TRIAL: NCT03686800
Title: The Comfort and Adherence of Rivelin® Plain Patches in Vulva Lichen Sclerosus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermtreat (Industry)
Collaborators: Larix A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DT-001-R-002
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: VLS
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivelin® plain patches (Experimental): This is an open label study with the objectives to establish information on adhesion time, tolerability and usability of Rivelin® plain patches when applied to VLS lesions. Furthermore, the design of the Rivelin® plain patch will also be evaluated.
  Interventions: Device: Rivelin® plain patches

INTERVENTIONS:
Device: Rivelin® plain patches — The comfort and adherence of Rivelin® plain patches in Vulva Lichen Sclerosus patients

SUMMARY:
This explorative investigation will assess the adhesion and tolerability of the Rivelin® plain patch when applied directly on lesions in subjects with Vulvar Lichen Sclerosus (VLS).

DETAILED DESCRIPTION:
The Rivelin® plain patch works by forming a protective barrier over a lesion, protecting it from further irritation and thus providing pain relief in much the same way as the adhesive pastes and films that are available to treat VLS. However, the adhesion/protection time of the Rivelin® plain patch is expected to be longer compared to current treatment with bioadhesive agents, thereby potentially increasing the pain free period for the subject.

This study is undertaken to gather information covering adhesion time and tolerability of the Rivelin® plain patch on areas affected by VLS. Since protecting a lesion with a physical barrier could reduce the sensation of pain caused by normal function, this investigation will also explore subject experienced pain and/or symptom relief during use of the patch for further development.

ELIGIBILITY:
Inclusion Criteria:

1. Women (≥ 18 years) diagnosed with VLS
2. Has received written and oral study information
3. Has given her written consent to study participation

Exclusion Criteria:

1. Pregnant
2. Menstruating at the time of patch application
3. Unable to communicate clearly with the examining doctors
4. Under the guardianship of another person or institution

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Adhesion time for Rivelin® plain patches | 2 days
  The proportion of successful applications of Rivelin® plain patches (defined as an adhesion time ≥ 30 min); separate summaries for morning and evening applications

SECONDARY OUTCOMES:
Adverse Events | 2 days
  Frequency and intensity of adverse events (AEs) and adverse device effects (ADEs) collected during the investigation
Ability to apply patches correctly | 2 days
  Study staff reported observation on subject's ability to apply patches correctly
Understanding of the Instructions for use leaflet | 2 days
  Subject reported outcome on the understanding of the Instructions for use leaflet
Visual analogue scale (VAS) scores | 2 days
  Visual analogue scale (VAS) scores for discomfort, pain, itching and burning prior to applying the first patch, at 2 hours after application (or when the first patch detaches) and on day 2
Optimising the design of the patch | 2 days
  Subject responses towards optimising the design of the patch

CONTACTS AND LOCATIONS:
Overall Officials: Gregor B.E. Jemec, MD, Principal Investigator — Zealand University Hospital, Dermatology dpt.
Locations (1):
- Zealand University Hospital, Dermatology dpt., Roskilde, Denmark